CLINICAL TRIAL: NCT03587558
Title: Effects of Carvedilol on Suppressing the Premature Ventricular Complex/Ventricular Tachycardia From Outflow Tract
Acronym: FOREVER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Collaborators: Chong Kun Dang Pharmaceutical Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-07-022
Record Dates: First submitted 2018-07-02; First posted 2018-07-16 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Ventricular Premature Complexes; Outflow Tract; Carvedilol
Keywords: carvedilol; SOICR; triggered activity; outflow tract PVC/VT
MeSH Terms: conditions — Ventricular Premature Complexes | interventions — Carvedilol; Flecainide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carvedilol group (Experimental): Patients in this group are taking carvedilol to inhibit outflow tract PVC/VT. Dilatrend® sustained release form of Chong Kun Dang Pharmaceutical will be used (initial dose: 8 mg sustained release form). Outpatient follow-up will be performed every 2 weeks and the dose is increased from the initial dose to a maximal tolerable dose, at the discretion of the investigator.
  Interventions: Drug: Carvedilol
- Flecainide group (Active Comparator): Patients in this group are taking flecainide to inhibit outflow tract PVC/VT. Tambocor® of JW Pharmaceutical will be used. Outpatient follow-up will be performed every 2 weeks and the dose is increased from the initial dose to a maximal tolerable dose, at the discretion of the investigator.
  Interventions: Drug: Flecainide

INTERVENTIONS:
Drug: Carvedilol — Patients in this group are taking carvedilol to inhibit outflow tract PVC/VT.
  Other Names: Dilatrend
  Arms: Carvedilol group
Drug: Flecainide — Patients in this group are taking flecainide to inhibit outflow tract PVC/VT.
  Other Names: Tambocor
  Arms: Flecainide group

SUMMARY:
Carvedilol is known to be effective in reducing ventricular arrhythmias and mortality in patients with heart failure. It is suggested that one of the mechanisms is its ability to block store overload-induced Calcium release which activates spontaneous calcium release by Ryanodine receptors. Ventricular outflow tract tachyarrhythmia is known to be associated with calcium overload due to activation of Ryanodine receptors. The aim of this study is to evaluate the efficacy of Carvedilol on premature ventricular complex(PVC)/ventricular tachycardia(VT) originating from outflow tract.

DETAILED DESCRIPTION:
Carvedilol is one of the third-generation beta-blockers effective in reducing ventricular arrhythmias and mortality in patients with heart failure. Antioxidative and alpha - blocking effects, along with nonselective beta - blockade, have been described as a mechanism of effect in various diseases.

The antiarrhythmic effect of carvedilol inhibiting atrial fibrillation or ventricular arrhythmia has been reported, but its mechanism is not yet clear. Among them, inhibition of store overload-induced Ca2+ release (SOICR) is suggested as an antiarrhythmic mechanism of carvedilol.

Stimulation of the beta receptor leads to the entry of calcium into the sarcoplasmic reticulum (SR) by opening the L-type calcium channel. The influx of calcium through the L-type calcium channel also increases the calcium release through the Ryanodine receptor (RyR) in the sarcoplasmic reticulum. This is called Ca-induced Ca release and is known as a normal physiological response. However, when calcium overload in the myofibrillar body occurs, spontaneous calcium release, known as SOICR, can occur through RyR, which can make triggered activity by inducing Na+/Ca2+ exchanger present in myocardium, leading to severe arrhythmia. Among several beta-blockers, only carvedilol has been known as a drug that can directly inhibit SOICR in combination with beta-blockade effect.

Ventricular tachyarrhythmia originating from the ventricular outflow tract is an arrhythmia occurring in a patient with normal cardiac function. The mechanism of the arrhythmia is known to be triggered activity which is caused by activation of RyR due to increased cyclic adenosine monophasphate, resulting in calcium overload, eventually causing activation of Na+/Ca2+ exchanger. The aim of this study is to evaluate the efficacy of Carvedilol on PVC/VT originating from outflow tract.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ventricular premature complexes/ventricular tachycardias originating from ventricular outflow tract confirmed on the 12-lead surface ECG
* Patients with PVC burden of 5% or more in 24-hour Holter monitoring
* Patients with normal left ventricular function

  * left ventricular ejection fraction ≥50%
* Patients without structural heart disease

Exclusion Criteria:

* Pregnant, trying to become pregnant or breast feeding
* History of bronchial asthma
* History of coronary arterial disease

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2017-09-05 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
PVC burden | 3 months after reaching the maximum tolerated dose
  Percentage of PVC/VT beat out of 24 hour total heart beat in Holter monitoring

SECONDARY OUTCOMES:
Symptom assessment scale | 3 months after reaching the maximum tolerated dose
  questionnaire for PVC/VT symptoms using symptom assessment scale (Min 0 to Max 100)
Side effect of drugs | 3 months after reaching the maximum tolerated dose
  Difference in occurrence of side effects of each drug

CONTACTS AND LOCATIONS:
Overall Officials: Seongwook Han, M.D., Ph.D., Study Chair — Keimyung University Dongsan Medical Center
Locations (11):
- South Korea (11):
  - Keimyung University Dongsan Medical Center, Daegu
  - Division of Cardiology, Department of Internal Medicine, Kyungpook National University Hospital, Daegu
  - Division of Cardiology, Department of Internal Medicine, Yeungnam University Hospital, Daegu
  - Division of Cardiology, Department of Internal Medicine, Daegu Catholic University Medical Center, Daegu
  - Chonnam National University Hospital, Gwangju
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Cardiovascular Hospital, Seoul
  - Seoul Asan Medical Center, Seoul
  - Seoul Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external independent Review Panel. Requestors will be required to sign a Data Access Agreement.